CLINICAL TRIAL: NCT00528671
Title: Effects of Very Low Dose Oral Anticoagulation on Thromboembolism and Bleeding Events in Patients With Mechanical Heart Valve Replacement
Brief Title: Very Low Dose Oral Anticoagulation and Thromboembolic and Bleeding Complications
Acronym: ESCAT III
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Collaborators: Klinikum Ludwigshafen (Other); University of Kiel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Mechanical Heart Valve Recipients
Keywords: phenprocoumon; INR self-management; mechanical heart valve replacement; bleeding; thromboembolism
MeSH Terms: conditions — Hemorrhage; Thromboembolism | interventions — Phenprocoumon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Low dose oral anticoagulation, INR self-management once a week
  Interventions: Drug: phenprocoumon
- B (Active Comparator): very low dose oral anticoagulation, INR self-management once a week
  Interventions: Drug: phenprocoumon
- C (Experimental): very low dose oral anticoagulation, INR self-management twice a week
  Interventions: Drug: phenprocoumon

INTERVENTIONS:
Drug: phenprocoumon — The daily phenprocoumon dose administered should achieve an international normalized ratio (INR) of 1.8 - 2.8 for aortic valve recipients and 2.5 - 3.5 for mitral or double valve recipients, INR-self management once a week
  Arms: A
Drug: phenprocoumon — The daily phenprocoumon dose administered should achieve an international normalized ratio (INR) of 1.6-2.1 for aortic valve recipients and 2.0 - 2.5 for mitral or double valve recipients, INR self management once a week
  Arms: B
Drug: phenprocoumon — The daily phenprocoumon dose administered should achieve an international normalized ratio (INR) of 1.6-2.1 for aortic valve recipients and 2.0 - 2.5 for mitral or double valve recipients, INR self management twice a week
  Arms: C

SUMMARY:
We aim to investiagte whether very low dose self management of oral anticoagulation is superior to low dose oral anticoagulation in order to prevent bleeding events in patients undergoing mechanuical heart valve replacement.

DETAILED DESCRIPTION:
In mechanical heart valve recipients, self-management of oral anticoagulation can reduce the risk of developing thromboembolic events and improves long-term survival compared with international normalized ratio (INR) control by a general practitioner. Low-dose INR self-management (INR values of 1.8.-2.8 for aortic valve recipients and 2.5 - 3.5 for mitral or double valve recipients) does not increase the risk of thromboembolic events compared to conventional dose INR self-management. Even in patients with a low INR target range, however, the risk of bleeding events is still higher than the risk of thromboembolism. We therefore perform a prospective, randomized trial in 1,800 patients with mechanical heart valve replacement. During the first six postoperative months, low dose INR self-management will be performed by all patients (INR measurement once a week). Thereafter, 600 patients will continue with this treatment regimen, whereas the other 1,200 patients with perform very low dose oral anticoagulation. Out of these 1,200 patients, 600 will perform INR measurement once a week and 600 patients will perform INR measurement twice a week. Patients are followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical heart valve recipients

Exclusion Criteria:

* Contra-indication to phenprocoumon
* Ulcerous disease with bleeding tendency,
* Hypo- or hypercoagulability
* Dementia
* Missing informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1571 (Actual)
Dates: Start 2006-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Thromboembolic events, Bleeding events, Survival rates | 2 years

SECONDARY OUTCOMES:
INR values, Percent of INR values in the target range | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Koertke, MD, Principal Investigator — Institute of Applied Telemedicine, Heart and Diabetes Center North-Rhine Westfalia, 32545 Bad Oeynhausen, Germany
Locations (1):
- Heart and Diabetes Center NRW, Bad Oeynhausen, Germany

REFERENCES:
- [Background] Koertke H, Minami K, Boethig D, Breymann T, Seifert D, Wagner O, Atmacha N, Krian A, Ennker J, Taborski U, Klovekorn WP, Moosdorf R, Saggau W, Koerfer R. INR self-management permits lower anticoagulation levels after mechanical heart valve replacement. Circulation. 2003 Sep 9;108 Suppl 1:II75-8. doi: 10.1161/01.cir.0000089185.80318.3f. PMID 12970212
- [Background] Koertke H, Zittermann A, Wagner O, Koerfer R. Self-management of oral anticoagulation therapy improves long-term survival in patients with mechanical heart valve replacement. Ann Thorac Surg. 2007 Jan;83(1):24-9. doi: 10.1016/j.athoracsur.2006.08.036. PMID 17184625
- [Background] Koertke H, Zittermann A, Mommertz S, El-Arousy M, Litmathe J, Koerfer R. The Bad Oeynhausen concept of INR self-management. J Thromb Thrombolysis. 2005 Feb;19(1):25-31. doi: 10.1007/s11239-005-0937-1. PMID 15976964
- [Background] Koertke H, Zittermann A, Minami K, Tenderich G, Wagner O, El-Arousy M, Krian A, Ennker J, Taborski U, Klovekorn WP, Moosdorf R, Saggau W, Morshuis M, Koerfer J, Seifert D, Koerfer R. Low-dose international normalized ratio self-management: a promising tool to achieve low complication rates after mechanical heart valve replacement. Ann Thorac Surg. 2005 Jun;79(6):1909-14; discussion 1914. doi: 10.1016/j.athoracsur.2004.09.012. PMID 15919283